CLINICAL TRIAL: NCT05826587
Title: A Mobile-Health (mHealth) Fall Risk Prevention Intervention in Cardiac Rehabilitation: A Randomized Control Trial
Brief Title: Cardiac Rehabilitation Mobile-Health Fall Risk Prevention Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert Scales, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-001155
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Rehabilitation
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group of cardiac rehabilitation only (Active Comparator)
  Interventions: Behavioral: Cardiac Rehabilitation & Exercise Prescription; Other: Connected mHealth mobile application
- Intervention group of additional balance and muscle strength training (Experimental)
  Interventions: Behavioral: Home-based, m-Health Delivered Physical Function Training; Behavioral: Cardiac Rehabilitation & Exercise Prescription; Other: Connected mHealth mobile application

INTERVENTIONS:
Behavioral: Home-based, m-Health Delivered Physical Function Training — An individualized home exercise physical function training will be prescribed. This would include 5 balance training exercises and 1-2 upper and lower-body muscular conditioning exercises (i.e., wall push-up and chair stand) prescribed 3 days/week over the course of a 6-week period. Subjects will be assigned exercises from 1 of 3 different levels of exercise progression based on performance during the baseline muscular fitness assessment (functional chair stand and static chest throw).
  Arms: Intervention group of additional balance and muscle strength training
Behavioral: Cardiac Rehabilitation & Exercise Prescription — Standard, clinically indicated cardiac rehabilitation and exercise program. Approximately 30 to 40 minutes of aerobic exercise within a prescribed rating of perceived exertion (RPE 11-14) and/or target heart rate and approximately 15 to 20 minutes of both upper and lower body resistance exercise up to three times per week for up to at least 12 weeks. In addition, subjects are provided with home exercise instructions, and will be expected to exercise for 30 to 60 minutes at home.
Other: Connected mHealth mobile application — Mobile application that allows subjects to track their independent home exercise with the option of heart rate monitoring by connecting to an external heart rate monitoring device.

SUMMARY:
The purpose of this research is to see if taking part in a structured exercise plan that is designed to improve balance and muscle strength and one that can done at home helps to improve the ability to perform standard physical tasks, confidence in balance, and health-related quality-of-life

DETAILED DESCRIPTION:
Traditional cardiac rehabilitation programs typically prioritize aerobic exercise (e.g., walking, cycling, etc.) with much less emphasis on improving physical function and strength, which is very important in, for example, decreasing the risk of falling. Through this research, researchers will implement a comprehensive fall risk screening and physical function assessment supported with individualized therapeutic exercise(s). Researchers hope that this will decrease fall risk, enhance rehabilitation experience, and improve ability to perform tasks of daily living.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to and who undergo early outpatient CR irrespective of diagnosis will be eligible for the study.
* All participants must have access to a smart mobile device.

Exclusion Criteria:

* Advanced dementia.
* Wheelchair bound.
* Vision loss.
* Patients that underwent sternotomy within 12-weeks will be excluded from the upper body muscular strength/power assessment and associated upper body training. At the time of enrollment into CR, balance, upper body muscular fitness, and lower body muscular fitness will be assessed in each subject before they are randomized at a 1:1 allocation ratio into one of two parallel groups:
* Standard early outpatient center-based supervised CR only (control; CR); or
* Early outpatient center-based supervised CR plus individualized, home-based, m-Health delivered physical function training (experimental group; CR+PFt). Balance, upper body muscular fitness, and lower body muscular fitness and gait will be reassessed in each participant after 5-to-6 weeks of CR and again upon completion of the CR program. Patient reported measures of fall risk will be measured at baseline with the Stop Elderly Accidents, Deaths, and Injuries (STEADI) tool kit. Balance confidence, health-related quality of life, physical activity level, and functional capacity will be evaluated before and after CR and CR+PFt using the Activities-Specific Balance Confidence (ABC) Scale, the Dartmouth Primary Care Cooperative Information Project (COOP) charts, and the Duke Activity Status Index (DASI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported physical function | Baseline, approximately 7 to 14 weeks
  Measured using the Duke Activity Status Index (DASI) a self-reported questionnaire to subjectively measure physical activity level and functional capacity. The questionnaire includes twelve questions with each question weighted differently to assign a total score. Functional capacity is graded based on the total score (i.e., Good = DASI >31.95 or Poor = DASI <31.95).
Change in fall risk | Baseline, approximately 7 to 14 weeks
  Measured using the Stop Elderly Accidents, Deaths, and Injuries (STEADI) assessment component which consists of 12 closed-ended questions. A score >4 is considered at risk for falling.
Change in self-reported balance confidence | Baseline, approximately 7 to 14 weeks
  Measured using the Activities-Specific Balance Confidence Scale, a 16-item questionnaire that is scored with a Likert scale (0-100%). The subject is graded on level of confidence associated with fall risk while performing a range of daily activities with varying levels of difficulty. Higher scores greater confidence.
Change in health-related quality of life | Baseline, approximately 7 to 14 weeks
  Measured using the Dartmouth Primary Care Cooperative Information Project (COOP), a nine-question quality of life survey. There are nine categories including: physical condition, emotional condition, daily work, social activities, change in condition, overall condition, social support, quality of life and pain. Subjects will be graded with a total and sub-category score. Total scores range from 9-45 and a lower total score indicates a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Scales, PhD, MS, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials